CLINICAL TRIAL: NCT06168708
Title: The Safety and Efficacy of Addition of Gentamicin on Irrigation Fluid in Prevention of Post-Transurethral Resection of the Prostate Infectious Complications: A Prospective Randomized Double Blinded Placebo Controlled Pilot Trial.
Brief Title: The Safety and Efficacy of Addition of Gentamicin on Irrigation Fluid in Prevention of Post-Transurethral Resection of the Prostate Infectious Complications.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Zoeir, faculty of medicine, Tanta, ElGeish street, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35121/12/21
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Post-TURP Infectious Complications
MeSH Terms: interventions — Transurethral Resection of Prostate; Gentamicins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Garamicin group (Active Comparator): the participants in this arm will undergo TURP with addition of one ampoule of gentamicin 80 mg (2ml) /3L of irrigation solution (the first 9 Liters during resection and the first 6 Liters during post-operative irrigation)
  Interventions: Procedure: Transurethral resection of the prostate (TURP); Drug: Gentamicin
- control group (Placebo Comparator): the participants in this arm will undergo TURP with addition of normal saline (2 ml) on the irrigation solution (placebo).
  Interventions: Procedure: Transurethral resection of the prostate (TURP); Drug: normal saline

INTERVENTIONS:
Procedure: Transurethral resection of the prostate (TURP) — TURP with addition of gentamicin on irrigation fluid to reduce infectious complications
Drug: Gentamicin — gentamicin 80 mg (2ml) /3L of irrigation solution (the first 9 Liters during resection and the first 6 Liters during post-operative irrigation)
  Arms: Garamicin group
Drug: normal saline — normal saline (2 ml) on the irrigation solution (placebo)
  Arms: control group

SUMMARY:
The aim of this clinical study is to evaluate the safety and efficacy of addition of gentamicin on irrigation fluid during trans-urethral resection of the prostate (TURP) and its role in reduction of post-TURP infectious complications.

the participants will be randomly divided into two groups: Group A (gentamicin group) and group B (Placebo).

DETAILED DESCRIPTION:
220 patients scheduled for TURP for the management of urinary retention or LUTS will be included and divided into two groups; "Group A" includes 110 patients who will undergo TURP with addition of one ampoule of gentamicin 80 mg (2ml) /3L of irrigation solution (the first 9 Liters during resection and the first 6 Liters during post-operative irrigation) and "Group B" includes 110 patients who will undergo TURP with addition of normal saline (2 ml) as a placebo on the irrigation solution. Determination of Gentamicin in human serum using HPLC/UV after Chemical Derivatization will be done using the method of Barends et al (Barends, Brouwers, & Hulshoff, 1987). Both groups will be compared as regards the demographic data, post-operative pyuria and bacteruria (1 week after removal of urethral catheter), fever, and/or sepsis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with enlarged prostate presenting with LUTS or urine retention

Exclusion Criteria:

* Unfit patients
* Renal impairment
* active UTI
* urethral strictures

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-12-07 (Estimated); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-07-07 (Estimated)

PRIMARY OUTCOMES:
infectious complications | 1 week and 1 month after removal of urethral catheter
  Post-TURP pyuria and bacteruria

CONTACTS AND LOCATIONS:
Locations (1):
- Urolgy Departement, Faculty of Medicine, Tanta University, Tanta, Outside U.S./Canada, Egypt